CLINICAL TRIAL: NCT05596344
Title: A Single-center, Real-world Prospective Observational Study of the Incidence and Development of Anxiety and Depression in Patients With Malignant Tumors
Brief Title: Long-term Follow-up of Anxiety and Depression in Patients With Malignant Tumors
Status: Recruiting | Type: Observational
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Jiaqiang, associate chief physician, Henan Cancer Hospital
Other Study IDs: ZZUSC-16
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Malignant Tumor; Anxiety; Depression
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Depression | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Hospital Anxiety and Depression Scale — The basic information, anxiety and depression, treatment and prognosis of these patients were collected.

SUMMARY:
This study was a single-center prospective, real-world observational study with plans to enroll all eligible patients. The basic information, anxiety and depression, treatment and prognosis of these patients were collected.

DETAILED DESCRIPTION:
A total of 200 patients with malignant tumors will be enrolled in Henan Cancer Hospital. This study is a single-center prospective real-world observational study, and all eligible patients are planned to be enrolled. The basic information, anxiety and depression, treatment and prognosis of these patients were collected.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women of all ages are welcome.
2. Pathological diagnosis of malignant tumor in our hospital.
3. Received at least one hospitalization at this hospital.
4. The expected survival time is greater than 1 year.

Exclusion Criteria:

1.There was no pathological report of malignancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with malignant tumors diagnosed by pathology receiving inpatient treatment in Henan Cancer Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2032-11-30 (Estimated); Study Completion 2032-11-30 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety Depression Scale | Confirmed in 1 day
  Confirmed in 1 day
Hospital Anxiety Depression Scale | End of the treatment
  End of the treatment
Hospital Anxiety Depression Scale | The treatment ended 3 months later
  The treatment ended 3 months later
Hospital Anxiety Depression Scale | The treatment ended 6 months later
  The treatment ended 6 months later
Hospital Anxiety Depression Scale | The treatment ended one year later
  The treatment ended one year later
Hospital Anxiety Depression Scale | The treatment ended 2 years ago
  The treatment ended 2 years ago

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Bone and Soft Tissue ,Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No